CLINICAL TRIAL: NCT02817165
Title: Probiotics in the Prevention of Antibiotic-Associated Diarrhea in Hospitalized Children: a Randomized Trial
Brief Title: Probiotics for the Prevention of Antibiotic-Associated Diarrhea
Acronym: PAID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: The Hospital for Sick Children (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Patricia Parkin, Research Director, Senior Associate Scientist and Professor, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000052303
Record Dates: First submitted 2016-04-12; First posted 2016-06-29 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Acute Diarrhea
Keywords: Probiotics, diarrhea, antibiotic, children, hospital
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (BioK+) (Experimental): Children will receive 10-40 billion CFUs/day of Bio-K+ (Lactobacillus acidophilus CL1285, Lactobacillus casei LBC80R and Lactobacillus rhamnosus CLR2), with dose based on their weight. The product will be administered as a strawberry flavored tub of milk.
  Interventions: Dietary Supplement: Probiotic (BioK+)
- Placebo (Placebo Comparator): Strawberry flavored tub of milk, identical (taste, color, odor) to the active Bio-K+ treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic (BioK+) — Probiotic (BioK+) with 3 stains of Lactobacillus
  Arms: Probiotic (BioK+)
Other: Placebo — Strawberry flavored tub of milk, identical (taste, color, odor) to the active Bio-K+ treatment.
  Arms: Placebo

SUMMARY:
In North America, one of the most common reasons for hospitalization in previously healthy children is for the treatment of infections with antibiotics. This study will determine if, in previously healthy children hospitalized and prescribed intravenous (IV) antibiotics, the co-administration of a probiotic milk product containing good bacteria, is safe and effective for reducing AAD, as compared to a placebo (identical appearing milk product). This will be a two-center, randomized, masked, placebo-controlled clinical trial. The results of this study will help inform clinicians and families on the use of probiotics in the prevention of AAD, a common side effect of antibiotic use among hospitalized children.

DETAILED DESCRIPTION:
A two-centred randomized, multi-blind (i.e. patients, caregivers, data collectors, outcome assessors, data managers and analysts), placebo-controlled clinical trial intended to evaluate the efficacy and safety of Bio-K+ (Lactobacillus acidophilus CL1285, Lactobacillus casei LBC80R and Lactobacillus rhamnosus CLR2) in the prevention of AAD in hospitalized children 1 year to 17 years of age administered IV antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be children aged 1 year to 17 years admitted to the General Pediatric inpatient unit at The Hospital for Sick Children (Site 1) or McMaster Children's Hospital (Site 2).
2. Participants will be prescribed IV antibiotics with a planned duration of 1 or more days, and a total course of both IV and oral antibiotics, if applicable, of no more than 28 days.
3. Parent (if parent-report) or patient (if patient-report) is able to communicate in English (read, write, speak).

Exclusion Criteria:

1. Parental or patient (e.g. child > 12 years old) report of current diarrhea, diarrhea within the last week.
2. Lactose intolerance.
3. Allergies to strawberry, dried citrus pulp, or any other components of the study product.
4. Immuno-compromised patients or those on immunosuppressive agents (e.g. heart or kidney transplant, complex care, sickle cell disease, chemotherapy agents, oral prednisone).
5. Patients with known or potentially compromised gut integrity (e.g. short gut, Inflammatory Bowel Disease, Celiac disease, Irritable Bowel Syndrome, nasogastric, nasojejunal or gastrostomy tube).
6. Children with serious and/or unstable medical conditions (e.g. diabetes, cardiovascular, renal, lung, psychiatric illness, bleeding disorders, etc.).
7. Children admitted to a medical or surgical subspecialty unit.
8. Patients enrolled in another study.
9. Patients previously randomized to this study.
10. Patient is pregnant.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence of antibiotic-associated diarrhea (AAD) | 2 weeks after antibiotic + probiotic completion
  The investigators will employ a questionnaire addressing Pediatric Acute Diarrhea (qPAD), a measure of diarrhea involving the assessment of stool frequency and consistency for each bowel movement. To measure consistency, the qPAD contains a stool consistency classification system. Our registered sample size is based on pilot data from The Hospital for Sick Children indicating that the incidence of AAD is 33% (95% CI 23% to 43%) according to the qPAD. Given an estimated baseline AAD risk of 32.9% and a 48% relative risk reduction in AAD (Johnston et al, Cochrane Library, 2011), a randomized trial with 80% power and a 2-sided alpha of 0.05 comparing Bio-K+ with placebo would require a total sample size of 118 patients per group (236 total).
Incidence of antibiotic-associated diarrhea (AAD), global impression | 2 weeks after antibiotic + probiotic completion
  Given that parents have knowledge of the child's typical bowel movements per day, the investigators will also employ a Global Rating Scale for diarrhea (GRSd), using a 0 to 4 scale (0 = no diarrhea, 1 = mild diarrhea, 2 = moderate diarrhea, 3 = severe diarrhea, 4 = worse imaginable diarrhea). The investigators will ask participants to select values based on diarrhea severity, which is a combination of stool frequency and consistency over 24 hours. Our registered sample size is based on the incidence of AAD (33%; 95% CI 23% to 43%) according to the qPAD. However, the incidence of AAD according to GRSd is 23%, which corresponds to the lower bound of the 95% CI for the qPAD. The investigators are currently applying for additional peer-reviewed funds. If these funds are obtained the investigators will power the trial based GRSd, a more conservative AAD incidence (23%). The investigators will also power the trial for a smaller treatment effect (39% relative risk reduction).

SECONDARY OUTCOMES:
Severity of AAD | 2 weeks after antibiotic completion
  The investigators will assess severity using the qPAD and the investigators will employ definitions for diarrhea from the Canadian Nosocomial Infection Surveillance Program, modified for use in children, defined as: severe: ≥6 loose/unformed/liquid stools; moderate: ≥3 loose/unformed/liquid stools; mild: a change in stooling pattern to 1-2 loose/unformed/liquid stools daily (Gravel 2007). The investigators will classify severity according to the 24-hour period with the highest degree of severity.
Adverse events | 2 weeks after antibiotic completion
  Incidence of mild (e.g. self-resolving), moderate (e.g. those that warrant medical evaluation) and serious (e.g. those that warrant continued hospitalization) adverse events based on criteria adopted by the National Institute of Health common terminology criteria for adverse events (NIH severity) will be evaluated.
Duration of AAD | 2 weeks after antibiotic completion
  The investigators will measure duration of AAD using a definition of diarrhea resolution (diarrhea offset) developed based on a systematic review of 138 trials of Pediatric Acute Diarrhea, and Delphi consensus with a panel of experts in pediatrics, clinical gastroenterology and measurement (Johnston BC et al. Pediatrics 2010; Jul;126(1):e222-31; Johnston BC et al. Symposium Probio, Quebec City, Canada, 2015).
  For children up to 17 years of age, acute diarrhea typically lasts less than 7 days and not longer than 14 days and resolution is marked by
  1. production of 2 consecutive normal stools (i.e. "soft and formed" or "hard and formed") stool or;
  2. production of one normal stool followed by 12 hours with no stool production or;
  3. normal stool production (or no stool production) for a period of 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Parkin, MD, Principal Investigator — The Hospital for Sick Children; Gordon Guyatt, MD, Study Chair — McMaster University
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
To be determined.

REFERENCES:
- [Background] Johnston BC, Shamseer L, da Costa BR, Tsuyuki RT, Vohra S. Measurement issues in trials of pediatric acute diarrheal diseases: a systematic review. Pediatrics. 2010 Jul;126(1):e222-31. doi: 10.1542/peds.2009-3667. Epub 2010 Jun 21. PMID 20566617
- [Background] Johnston B, Pirrello D, Lytvyn L, Mahant S, Sherman P, Ship N, Parkin P. Prospective cohort study of antibiotic-associated diarrhea among hospitalized children. Symposium Probio, Quebec City, Canada. (October 29, 2015).
- [Background] Goldenberg JZ, Lytvyn L, Steurich J, Parkin P, Mahant S, Johnston BC. Probiotics for the prevention of pediatric antibiotic-associated diarrhea. Cochrane Database Syst Rev. 2015 Dec 22;(12):CD004827. doi: 10.1002/14651858.CD004827.pub4. PMID 26695080